CLINICAL TRIAL: NCT03660826
Title: A Randomized Phase II Study Comparing Single-Agent Olaparib, Single Agent Cediranib, and the Combinations of Cediranib/Olaparib, Olaparib/Durvalumab (MEDI4736), Cediranib/Durvalumab (MEDI4736), Olaparib/AZD5363 (Capivasertib) in Women With Recurrent, Persistent or Metastatic Endometrial Cancer. A Multi-Arm Trial for Women With Recurrent or Persistent Endometrial Cancer
Brief Title: Testing the Combination of Olaparib and Durvalumab, Cediranib and Durvalumab, Olaparib and Capivasertib, and Cediranib Alone in Recurrent or Refractory Endometrial Cancer Following the Earlier Phase of the Study That Tested Olaparib and Cediranib in Comparison to Cediranib Alone, and Olaparib Alone
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01672; NCI-2017-01672 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY012 (Other: NRG Oncology); NRG-GY012 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2018-09-06; First posted 2018-09-07 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Endometrioid Adenocarcinoma; Stage IV Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8
MeSH Terms: conditions — Carcinoma, Endometrioid; Carcinosarcoma | interventions — Specimen Handling; Fluid Therapy; Biopsy; capivasertib; cediranib; durvalumab; Immunoglobulin G; Disulfides; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm I (cediranib maleate_reference group 1) (Experimental): Patients in reference group 1 receive cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Arm II (olaparib) (Experimental): Patients receive olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm III (cediranib maleate, olaparib) (Experimental): Patients receive olaparib PO BID and cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm IV (olaparib, capivasertib) (Experimental): Patients receive olaparib PO BID on days 1-28 and capivasertib PO BID on days 1-4 each week. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Capivasertib; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm V (olaparib, durvalumab) (Experimental): Patients receive olaparib PO BID on days 1-28 and durvalumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib
- Arm VI (cediranib maleate, durvalumab) (Experimental): Patients receive cediranib maleate PO QD on days 1-5 each week and durvalumab IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Cediranib Maleate; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Arm VII (cediranib maleate_reference group 2) (Experimental): Patients in reference group 1 receive cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow aspiration and biopsy
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
  Arms: Arm I (cediranib maleate_reference group 1); Arm II (olaparib); Arm III (cediranib maleate, olaparib); Arm IV (olaparib, capivasertib); Arm V (olaparib, durvalumab); Arm VI (cediranib maleate, durvalumab)
Drug: Capivasertib — Given PO
  Other Names: AZD 5363; AZD-5363; AZD5363; Truqap
  Arms: Arm IV (olaparib, capivasertib)
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm I (cediranib maleate_reference group 1); Arm III (cediranib maleate, olaparib); Arm VI (cediranib maleate, durvalumab); Arm VII (cediranib maleate_reference group 2)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm V (olaparib, durvalumab); Arm VI (cediranib maleate, durvalumab)
Procedure: Echocardiography Test — Undergo Echo
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm II (olaparib); Arm III (cediranib maleate, olaparib); Arm IV (olaparib, capivasertib); Arm V (olaparib, durvalumab)

SUMMARY:
This phase II trial studies the effects of the combination of olaparib and durvalumab, cediranib and durvalumab, olaparib and capivasertib, and cediranib alone in treating patients with endometrial cancer that has come back (recurrent) or does not respond to treatment (refractory). Olaparib, cediranib, and capivasertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Durvalumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Testing the combinations may lower the chance of endometrial cancer growing or spreading compared to usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the efficacy of single-agent olaparib and the combination of olaparib and cediranib (and potentially other combination arms that may be added by subsequent amendment) versus single agent cediranib as measured by progression free survival (PFS), in patients with recurrent, persistent or metastatic endometrial cancer.

II. To compare the efficacy of the combination of olaparib and AZD5363 (capivasertib), and the combination of olaparib and durvalumab (MEDI4736), and the combination of cediranib and durvalumab (MEDI4736) versus single agent cediranib as measured by progression free survival (PFS), in patients with recurrent, persistent or metastatic endometrial cancer.

SECONDARY OBJECTIVES:

I. To compare the efficacy of single-agent olaparib and the combination of olaparib and cediranib (and potentially other combination arms that may be added by subsequent amendment) versus single-agent cediranib as measured by overall survival (OS) in patients with recurrent, persistent or metastatic endometrial cancer.

II. To compare the efficacy of the combination of olaparib and AZD5363 (capivasertib), and the combination of olaparib and durvalumab (MEDI4736), and the combination of cediranib and durvalumab (MEDI4736) versus single agent cediranib as measured by overall survival (OS), in patients with recurrent, persistent or metastatic endometrial cancer.

III. To compare the efficacy of single-agent olaparib and the combination of olaparib and cediranib (and potentially other combination arms may be added by subsequent amendment versus single-agent cediranib as measured by response rate in patients with recurrent, persistent or metastatic endometrial cancer.

IV. To compare the efficacy of the combination of olaparib and AZD5363 (capivasertib), and the combination of olaparib and durvalumab (MEDI4736), and the combination of cediranib and durvalumab (MEDI4736) versus single agent cediranib as measured by response rate in patients with recurrent, persistent or metastatic endometrial cancer.

V. To assess the safety and tolerability of single-agent cediranib, single-agent olaparib, and the combination of olaparib and cediranib (and potentially other combination arms may be added by subsequent amendment).

VI. To assess the safety and tolerability of the combination of olaparib and AZD5363 (capivasertib), and the combination of olaparib and durvalumab (MEDI4736), and the combination of cediranib and durvalumab (MEDI4736).

VII. To assess if mutations in deoxyribonucleic acid (DNA) homologous repair genes (assayed prior to all treatment and prior to the study treatment) are predictive of response to olaparib alone or in combination with cediranib. (Integrated Biomarker) VIII. To assess if markers of angiogenesis in serial plasma samples are associated with response to cediranib alone or in combination with olaparib. (Integrated Biomarker)

EXPLORATORY OBJECTIVE:

I. To compare the efficacy of the combination of olaparib and cediranib versus single agent olaparib as measured by PFS, response rate and OS, if and only if the combination is superior to the single-agent cediranib arm.

OUTLINE: Patients are randomized to 1 of 6 arms.

ARM I: Patients in reference group 1 receive cediranib maleate orally (PO) once daily (QD). Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, computed tomography (CT), echocardiography (Echo) or multigated acquisition scan (MUGA) on study.

ARM II: Patients receive olaparib PO twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

ARM III: Patients receive olaparib PO BID and cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

ARM IV: Patients receive olaparib PO BID on days 1-28 and capivasertib PO BID on days 1-4 each week. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

ARM V: Patients receive olaparib PO BID on days 1-28 and durvalumab intravenously (IV) on day 1. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

ARM VI: Patients receive cediranib maleate PO QD on days 1-5 each week and durvalumab IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

ARM VII: Patients in reference group 1 receive cediranib maleate PO QD during 08/16/2021 - 06/28/2023). Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required; patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.); NOTE: clear cell histology is excluded.
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or non-measurable (detectable) disease

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI; patients with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
  * Non-measurable (detectable) disease in a patient is defined in this protocol as one who does not have measurable disease but has at least one of the following conditions:

    * Ascites and/or pleural effusion attributed to tumor;
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen.
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition: cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa; Note: patients on this non-cytotoxic study are allowed to receive one additional cytotoxic chemotherapy regimen for management of recurrent or persistent disease, as defined above; however, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy.
* Patients may have received non cytotoxic therapy including immunotherapy (1 prior line in either upfront or recurrent setting) but excluding cediranib, olaparib, AZD5363 (capivasertib), durvalumab (MEDI4736), or the combination of lenvatinib and pembrolizumab for the management of recurrent or persistent disease; prior hormonal therapy is allowed; hormonal therapy for grade 1 endometrial cancers with low volume or indolent disease is encouraged.
* Bevacizumab, or one course of single-agent immune-checkpoint therapy, excluding durvalumab (MEDI4736), is permitted prior to enrollment on this trial.
* Body weight > 30 kg.
* Age >= 18.
* The trial is open to females only (including women with an intact uterus with uterine cancer); fertile females of childbearing potential need to agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after study treatment discontinuation, and have a negative serum or urine pregnancy test within 3 days prior to the start of study treatment.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2 (Karnofsky >= 60%) within 7 days prior to registration; patients should have no deterioration over the previous two weeks.
* Hemoglobin >= 10 mg/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study drug).
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study drug).
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 28 days prior to administration of study drug).
* Patients must have creatinine clearance estimated of >= 51 mL/min using the Cockcroft Gault equation or based on a 24-hour urine test (within 28 days prior to administration of study drug).
* Serum bilirubin =< 1.5 X upper limit of normal (ULN) (within 28 days prior to administration of study drug).
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (within 28 days prior to administration of study drug).
* Urinalysis (dipstick) =< 1+ proteinuria OR urine protein creatinine ratio (UPCR) < 1 (within 28 days prior to administration of study drug).
* Patients must be able to swallow and retain oral medications and without gastrointestinal illnesses that would preclude absorption of cediranib, olaparib, or AZD5363 (capivasertib).
* Patients must have adequately controlled blood pressure (BP), with a BP no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility; patients must have a BP of =< 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to starting study; patients with hypertension may be managed with up to a maximum of three antihypertensive medications; it is strongly recommended that patients who are on three antihypertensive medications be followed by a cardiologist or blood pressure specialist for management of blood pressure while on protocol.

  * Note: Patients must be willing and able to check and record daily blood pressure readings.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry.
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to start of investigational products (IPs); postmenopausal is defined as:

  * Age >= 60 years, or
  * Age < 60 with any one or more of the conditions below:

    * Amenorrheic for >= 1 year in the absence of chemotherapy and/or hormonal treatments,
    * Luteinizing hormone and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range
    * Radiation-induced oophorectomy with last menses > 1 year ago,
    * Chemotherapy-induced menopause with > 1 year interval since last menses,
    * Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Patients must have a life expectancy of greater than 16 weeks.
* Patients with a previous diagnosis of immune or inflammatory colitis or chronic diarrhea > 1 month without immune or inflammatory colitis are eligible with adequately controlled colitis (no diarrhea greater than grade 1 for at least 28 days) and in the absence of symptoms related to colonic dysfunction; patients who required steroids for prior immune related colitis are not eligible.
* Females of child-bearing potential should use two forms of highly reliable methods of contraception from the time of screening until 4 weeks after discontinuing study treatment.

  * Acceptable methods of contraception include:

    * Established use of oral, injected or implanted hormonal methods of contraception.
    * Placement of an intrauterine device or intrauterine system.
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
    * True abstinence (i.e., not engaging in sexual activity for the total duration of study treatment and the treatment washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control).
    * Bilateral tubal occlusion or salpingectomy
  * Acceptable non-hormonal birth control methods include:

    * Total/True abstinence: When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle; this must continue for the total duration of the trial and for at least 1 month after the last dose of study drug <<for 3 months after last dose for male patients>>. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, or declaration of abstinence solely for the duration of a trial) and withdrawal are not acceptable methods of contraception]
    * Vasectomised sexual partner PLUS male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia.
    * Tubal occlusion PLUS male condom
    * Intrauterine device (IUD) PLUS male condom. Provided coils are copper-banded.
  * Acceptable hormonal methods:

    * Normal and low dose combined oral pills PLUS male condom.
    * Cerazette (desogestrel) PLUS male condom. Cerazette is currently the only highly efficacious progesterone-based pill.
    * Hormonal shot or injection (e.g., Depo-Provera) PLUS male condom.
    * Etonogestrel implants (e.g., Implanon, Norplant) PLUS male condom.
    * Norelgestromin/EE transdermal system PLUS male condom
    * Intrauterine system [IUS] device (e.g., levonorgestrel releasing IUS -Mirena) PLUS male condom.
    * Intravaginal device (e.g., EE and etonogestrel) PLUS male condom.

Exclusion Criteria:

* Prior enrollment into a clinical trial including cediranib or olaparib; Note: prior bevacizumab is not an exclusion criterion.
* Prior enrollment into a clinical trial including cediranib, olaparib, AZD5363 (capivasertib), durvalumab (MEDI4736), or the combination of lenvatinib and pembrolizumab. Note: Prior bevacizumab or single-agent immune checkpoint blockade, excluding durvalumab (MEDI4736), is not an exclusion criterion.
* Prior chemotherapy, endocrine therapy, radiotherapy, or investigational agents within 4 weeks.
* More than one prior line of treatment with immune checkpoint blockade therapy.
* Current signs/symptoms of bowel obstruction and/or signs/symptoms of bowel obstruction within the preceding 3 months.
* History of gastrointestinal perforation; patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula.
* Uncontrolled intercurrent illness including, but not limited to known ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or psychiatric illness/social situations that would limit compliance with study requirements.
* Concomitant use of known strong cytochrome (CYP) 3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil); the required washout period prior to starting study treatments is 2 weeks for strong inhibitors, and at least 1 week for moderate inhibitors.
* Concomitant use of potent inhibitors or inducers of CYP3A4 within 2 weeks before the start of study treatment (3 weeks for St John's wort), or sensitive substrates of CYP3A4, CYP2C9 and/or CYP2D6 with a narrow therapeutic window within 1 week before the start of study treatment. Concomitant use of drugs known to prolong the QT interval within 5 half-lives of the first dose of study treatment.
* Pregnant women are excluded from this study because cediranib and olaparib are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with cediranib and olaparib, breastfeeding should be discontinued if the mother is treated with cediranib or olaparib; these potential risks may also apply to other agents used in this study; for women of childbearing capacity a negative pregnancy test is required.
* Known human immunodeficiency virus (HIV)-positive individuals are ineligible because of the potential for pharmacokinetic interactions between many anti-HIV drugs and cediranib, olaparib, and/or AZD5363 (capivasertib); in addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Known active hepatitis B or hepatitis C infection on antiviral treatment.
* Prior history of stroke or transient ischemic attack within the last 6 months.
* Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) per institutional guidelines, or < 55%, if threshold for normal not otherwise specified by institutional guidelines, for patients with the following risk factors:

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * Prior central thoracic radiation therapy (RT), including exposure of heart to therapeutic doses of ionizing RT
  * History of myocardial infarction within 6-12 months prior to start of IPs
  * Prior history of other significant impaired cardiac function.
* Patients with any of the following:

  * History of myocardial infarction within 6 months prior to starting treatment
  * Unstable angina
  * Resting electrocardiogram (ECG) with clinically significant abnormal findings or with corrected QT interval (QTc) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
  * New York Heart Association functional classification of III or IV.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Major surgical procedure within 4 weeks prior to starting treatment; patients must have recovered from any effects of any major surgery and surgical wound should have healed prior to starting treatment.
* History of intra-abdominal abscess within 3 months prior to starting treatment.
* Patients may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments.
* No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUBCT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).
* Patients with myelodysplastic syndrome (MDS)/treatment-related acute myeloid leukemia (t-AML) or with features suggestive of MDS/AML.
* Central nervous system metastases:

  * Symptomatic uncontrolled brain metastases requiring corticosteroid treatment; history of spinal cord compression unless after definitive treatment the patient has clinically stable disease (SD) for at least 28 days prior to starting IPs; in the absence of these features and in an asymptomatic patient a scan to confirm the absence of brain metastases is not required.
* Other malignancy within the last 5 years except for:

  * Curatively treated basal cell or squamous cell carcinoma of skin; in situ cancer of the cervix, ductal carcinoma in situ of the breast or stage 1, grade 1 endometrial carcinoma
  * Curatively treated other solid tumors including lymphomas (without bone marrow involvement) with no evidence of disease for >= 5 years prior to start of IPs.
* Persisting >= grade 2 Common Terminology Criteria for Adverse Events (CTCAE) toxicity (except alopecia and grade 2 peripheral neuropathy) from previous anti-cancer treatment(s).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib, olaparib, AZD5363 (capivasertib), or durvalumab (MEDI4736).
* Pneumonitis or moderate-severe pre-existing pulmonary disease.
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days of enrollment.

  * Premedication with steroids for CT scan contrast is allowed.
  * Inhaled or topical corticosteroids are allowed.
  * The use of mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
  * The use of physiologic doses of corticosteroids may be approved after consultation with the study chair.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. This includes, but is not limited to, patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease.
* Patients with vitiligo, endocrine deficiencies including type I diabetes mellitus, thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible.
* Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2026-01-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Helen J Mackay, Principal Investigator — NRG Oncology
Locations (764):
- United States (763):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Providence Queen of The Valley, Napa, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Bradenton Cancer Center, Bradenton, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Florida Cancer Specialists - Venice Island, Venice, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Carle BroMenn Outpatient Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Baptist Health Richmond, Richmond, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rimel BJ, Enserro D, Bender DP, Jackson CG, Tan A, Alluri N, Borowsky M, Moroney J, Hendrickson AW, Backes F, Swisher E, Powell M, MacKay H. NRG-GY012: Randomized phase 2 study comparing olaparib, cediranib, and the combination of cediranib/olaparib in women with recurrent, persistent, or metastatic endometrial cancer. Cancer. 2024 Apr 15;130(8):1234-1245. doi: 10.1002/cncr.35151. Epub 2023 Dec 21. PMID 38127487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial first activated on 09/04/2018 with reporting groups 1-3. It closed to accrual for reporting groups 1-3 on 06/17/2019. It reopened to accrual for reporting groups 4-7 on 08/16/2021. It closed to accrual for reporting groups 4-7 on 06/28/2023.
Groups:
- Arm I (Cediranib maleate_Reference Group 1): Patients randomized to Cedinarib reference arm during the recruitment period (09/04/2018-06/17/2019). Patients receive Cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
- Arm II (Olaparib): Patients receive olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
  Olaparib: Given PO
- Arm III (Cediranib Maleate, Olaparib): Patients receive olaparib PO BID and cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
  Olaparib: Given PO
- Arm IV (Olaparib, Capivasertib): Patients receive olaparib PO BID on days 1-28 and capivasertib PO BID on days 1-4 each week. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Capivasertib: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
  Olaparib: Given PO
- Arm V (Olaparib, Durvalumab): Patients receive olaparib PO BID on days 1-28 and durvalumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Computed Tomography: Undergo CT scan
  Durvalumab: Given IV
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
  Olaparib: Given PO
- Arm VI (Cediranib Maleate, Durvalumab): Patients receive cediranib maleate PO QD on days 1-5 each week and durvalumab IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Durvalumab: Given IV
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
- Arm VII (Cediranib maleate_Reference Group 2): Patients randomized to Cedinarib reference arm during the recruitment period (08/16/2021-06/28/2023).
  Patients receive cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUG
Period: Overall Study
Arm/Group | Arm I (Cediranib maleate_Reference Group 1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Reference Group 2)
Started | 40 | 40 | 40 | 42 | 42 | 43 | 41
Completed | 40 | 40 | 40 | 42 | 42 | 43 | 41
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Cediranib maleate_Group1): Patients randomized to Cedinarib reference arm during the recruitment period (09/04/2018-06/17/2019). Patients receive Cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
- Arm VII (Cediranib maleate_Group2): Patients randomized to Cedinarib reference arm during the recruitment period (08/16/2021-06/28/2023).
  Patients receive cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
- Total: Total of all reporting groups
Arm/Group | Arm I (Cediranib maleate_Group1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Group2) | Total
Number analyzed (Participants) | 40 | 40 | 40 | 42 | 42 | 43 | 41 | 288
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  40-49 years | 5 | 0 | 3 | 1 | 4 | 2 | 3 | 18
  50-59 years | 5 | 2 | 2 | 1 | 5 | 6 | 3 | 24
  60-69 years | 20 | 24 | 25 | 24 | 23 | 21 | 20 | 157
  70-79 years | 10 | 13 | 10 | 14 | 7 | 12 | 12 | 78
  80-89 years | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 40 | 42 | 42 | 43 | 41 | 288
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 9
  Not Hispanic or Latino | 40 | 39 | 37 | 41 | 38 | 39 | 37 | 271
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 2 | 2 | 3 | 1 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 4 | 5 | 4 | 8 | 5 | 36
  White | 34 | 31 | 32 | 34 | 33 | 31 | 27 | 222
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 2 | 1 | 2 | 3 | 3 | 14
Prior Immunotherapy [Count of Participants; unit: Participants]
  No | 36 | 38 | 35 | 29 | 29 | 29 | 28 | 224
  Yes | 4 | 2 | 5 | 13 | 13 | 14 | 13 | 64
Histology [Count of Participants; unit: Participants]
  Serous | 15 | 16 | 16 | 17 | 18 | 13 | 18 | 113
  Endometrioid, Grade 1 | 6 | 2 | 7 | 5 | 3 | 9 | 7 | 39
  Endometrioid, Grade 2 | 9 | 6 | 8 | 11 | 11 | 10 | 6 | 61
  Endometrioid, Grade 3 | 4 | 11 | 5 | 6 | 6 | 10 | 8 | 50
  Other | 6 | 5 | 4 | 3 | 4 | 1 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the date of study enrollment to the investigator-determined date of progression or death due to any cause, whichever occurs first. For individuals who are alive and progression-free, the censored time at risk will be defined as the time from the study enrollment date to the date of the patient's last radiographic disease assessment.
Time Frame: Scans were done every 8 weeks for the first year and then every 12 weeks thereafter until disease progression. Vital status was assessed every 3 months for 2 years and then every 6 months for 3 years (5-years total).
Population: All patients randomized (Intent-to-Treat).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm VII (Cediranib maleate_Reference Group 2): Patients randomized to Cedinarib reference arm during the recruitment period (08/16/2021-06/28/2023).
  Patients receive cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
Arm/Group | Arm I (Cediranib maleate_Reference Group 1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Reference Group 2)
Number analyzed (Participants) | 40 | 40 | 40 | 42 | 42 | 43 | 41
Months | 3.8 [3.0 to 5.4] | 2.0 [1.8 to 4.7] | 5.5 [3.7 to 8.3] | 5.6 [2.6 to 6.0] | 3.7 [2.2 to 4.9] | 6.0 [3.8 to 7.8] | 4.1 [3.0 to 7.0]
Statistical Analysis 1: Comparison: Arm I (Cediranib maleate_Reference Group 1) vs Arm II (Olaparib); Test type: Superiority; p = 0.93, Log Rank — Comparing Arm II vs Arm I (reference group); Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.91 to 2.30]; Comparing Arm II vs Arm I (reference group)
Statistical Analysis 2: Comparison: Arm I (Cediranib maleate_Reference Group 1) vs Arm III (Cediranib Maleate, Olaparib); Comparing Arm III vs Arm I; Test type: Superiority; p = 0.06, Log Rank; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.43 to 1.14]
Statistical Analysis 3: Comparison: Arm IV (Olaparib, Capivasertib) vs Arm VII (Cediranib maleate_Reference Group 2); Comparing Arm IV vs Arm VII; Test type: Superiority; p = 0.62, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.67 to 1.70]
Statistical Analysis 4: Comparison: Arm V (Olaparib, Durvalumab) vs Arm VII (Cediranib maleate_Reference Group 2); Comparing Arm V vs Arm VII; Test type: Superiority; p = 0.36, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.58 to 1.46]
Statistical Analysis 5: Comparison: Arm VI (Cediranib Maleate, Durvalumab) vs Arm VII (Cediranib maleate_Reference Group 2); Comparing Arm VI vs VII; Test type: Superiority; p = 0.14, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.49 to 1.25]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of study enrollment to the date of death regardless of cause. For those individuals who have no death reported at the time of the analysis, the censored time at risk will be assessed from the date of study enrollment to the date that the patient was last contacted and known to be alive.
Time Frame: Vital status was assessed every 3 months for 2 years and then every 6 months for 3 years (5-years total).
Population: All patients randomized (Intent-to-Treat)
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm I (Cediranib maleate_Referenc Group 1): Patients randomized to Cedinarib reference arm during the recruitment period (09/04/2018-06/17/2019). Patients receive Cediranib maleate PO QD. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy, CT, Echo or MUGA on study.
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspirate: Undergo bone marrow aspiration and biopsy
  Bone Marrow Biopsy: Undergo bone marrow aspiration and biopsy
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT scan
  Echocardiography: Undergo Echo
  Multigated Acquisition Scan: Undergo MUGA
Arm/Group | Arm I (Cediranib maleate_Referenc Group 1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Reference Group 2)
Number analyzed (Participants) | 40 | 40 | 40 | 42 | 42 | 43 | 41
Months | 12.4 [7.5 to 22.9] | 13.4 [6.5 to 19.5] | 17.6 [9.3 to 21.2] | 16.9 [9.3 to 20.3] | 14.0 [10.4 to 20.3] | 22.6 [13.1 to NA] — The number of events was not sufficient for the estimation of this parameter (i.e. upper limit of the CI) | 16.6 [8.5 to 20.6]

3. Secondary Outcome: Objective Tumor Response
Description: Objective tumor response was assessed in patients with measurable disease by the site investigator using RECIST v1.1. Patients with complete or partial tumor response were considered to have a response.
Time Frame: Scans were done every 8 weeks for the first year; then every 12 weeks thereafter until disease progression is confirmed or up to 33 months.
Population: All patients who are eligible for response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cediranib maleate_Group1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Group2)
Number analyzed (Participants) | 29 | 32 | 35 | 38 | 32 | 34 | 30
Participants | 7 | 4 | 11 | 8 | 11 | 16 | 6

4. Secondary Outcome: Incidence of Adverse Events
Description: The number of patients who reported at least a grade 3 adverse event were assessed in those who initiated treatment.
Time Frame: Toxicity was assessed every other week for the first 8 weeks of study therapy and every 8 weeks after the completion or termination of study therapy up to 50 months.
Population: Patients who initiated assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cediranib maleate_Group1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Group2)
Number analyzed (Participants) | 39 | 40 | 39 | 42 | 42 | 42 | 37
Participants | 28 | 19 | 31 | 24 | 21 | 31 | 28

5. Other Pre Specified Outcome: Mutations in Deoxyribonucleic Acid (DNA) Homologous Repair Genes
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Markers of Angiogenesis in Serial Plasma Samples
Description: Will assess if markers of angiogenesis in serial plasma samples are associated with response to cediranib alone or in combination with olaparib.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Toxicity was assessed every other week for the first 8 weeks of study therapy and every 8 weeks after the completion or termination of study therapy. Median follow-up was 22 months.
Description: Patients randomized were included for the all-cause mortality summary. Patients randomized and also initiated treatment were included for the AE/SAE summary.
Arm/Group | Arm I (Cediranib maleate_Reference Group 1) | Arm II (Olaparib) | Arm III (Cediranib Maleate, Olaparib) | Arm IV (Olaparib, Capivasertib) | Arm V (Olaparib, Durvalumab) | Arm VI (Cediranib Maleate, Durvalumab) | Arm VII (Cediranib maleate_Reference Group 2)
All-Cause Mortality (participants affected / at risk) | 23/40 | 26/40 | 20/40 | 27/42 | 28/42 | 21/43 | 27/41
Serious Adverse Events (participants affected / at risk) | 17/39 | 12/40 | 19/39 | 11/42 | 16/42 | 13/42 | 19/37
Other Adverse Events (participants affected / at risk) | 38/39 | 40/40 | 39/39 | 41/42 | 42/42 | 40/42 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cediranib maleate_Reference Group 1) (N=39) | Arm II (Olaparib) (N=40) | Arm III (Cediranib Maleate, Olaparib) (N=39) | Arm IV (Olaparib, Capivasertib) (N=42) | Arm V (Olaparib, Durvalumab) (N=42) | Arm VI (Cediranib Maleate, Durvalumab) (N=42) | Arm VII (Cediranib maleate_Reference Group 2) (N=37)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 2
Colonic Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
General Disorders And Administration Site Conditio (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Edema Limbs (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death Nos (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight Loss (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Ggt Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft Tissue Necrosis Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Weakness Left-Sided (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cediranib maleate_Reference Group 1) (N=39) | Arm II (Olaparib) (N=40) | Arm III (Cediranib Maleate, Olaparib) (N=39) | Arm IV (Olaparib, Capivasertib) (N=42) | Arm V (Olaparib, Durvalumab) (N=42) | Arm VI (Cediranib Maleate, Durvalumab) (N=42) | Arm VII (Cediranib maleate_Reference Group 2) (N=37)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 12 | 27 | 10 | 24 | 21 | 11 | 5
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 1
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0 | 1 | 1 | 2
Cardiac Disorders - Other (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 3
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Heart Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hearing Impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endocrine Disorders - Other (Endocrine disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 0 | 1 | 0 | 0 | 5 | 3
Hypothyroidism (Endocrine disorders) | 10 | 1 | 11 | 2 | 1 | 12 | 18
Vision Decreased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Disorders - Other (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4
Flashing Lights (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blurred Vision (Eye disorders) | 2 | 1 | 2 | 1 | 3 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Watering Eyes (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 30 | 10 | 26 | 31 | 10 | 26 | 31
Dry Mouth (Gastrointestinal disorders) | 4 | 0 | 6 | 4 | 1 | 6 | 7
Constipation (Gastrointestinal disorders) | 9 | 9 | 11 | 10 | 11 | 14 | 12
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colonic Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 16 | 8 | 14 | 15 | 12 | 7 | 7
Stomach Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rectal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 3 | 1 | 3
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 22 | 24 | 28 | 29 | 20 | 18 | 25
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 1 | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 10 | 1 | 9 | 4 | 3 | 6 | 11
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 2 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 2 | 0 | 4 | 4 | 1 | 3 | 0
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Dysesthesia (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 2
Oral Pain (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 0 | 1 | 1
Anal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 13 | 8 | 10 | 9 | 11 | 14 | 12
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Belching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 0 | 4 | 1 | 4 | 2
Pain (General disorders) | 4 | 4 | 6 | 4 | 2 | 2 | 5
Malaise (General disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1
Flu Like Symptoms (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Fever (General disorders) | 4 | 2 | 1 | 5 | 1 | 4 | 1
General Disorders And Administration Site Conditio (General disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 1
Fatigue (General disorders) | 25 | 28 | 29 | 30 | 22 | 22 | 23
Gait Disturbance (General disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 1
Edema Trunk (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 3
Edema Limbs (General disorders) | 1 | 8 | 3 | 4 | 10 | 5 | 3
Edema Face (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Localized Edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Immune System Disorders - Other (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1
Wound Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vulval Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 7 | 4 | 5 | 4 | 7 | 5 | 7
Thrush (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 2 | 3
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 1 | 0
Shingles (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Rhinitis Infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papulopustular Rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 4 | 0 | 0 | 1 | 1 | 0 | 0
Infections And Infestations - Other (Infections and infestations) | 1 | 0 | 1 | 3 | 3 | 3 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes Simplex Reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1 | 0 | 2 | 0 | 3 | 1
Bronchial Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bladder Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0 | 2 | 3 | 1
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 4 | 3 | 0 | 1 | 2 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Weight Loss (Investigations) | 15 | 6 | 14 | 5 | 7 | 11 | 11
Weight Gain (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Thyroid Stimulating Hormone Increased (Investigations) | 6 | 0 | 6 | 3 | 4 | 5 | 7
Serum Amylase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Platelet Count Decreased (Investigations) | 5 | 4 | 8 | 6 | 6 | 3 | 7
Neutrophil Count Decreased (Investigations) | 3 | 5 | 5 | 4 | 7 | 1 | 5
Lymphocyte Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 3 | 3 | 7 | 12 | 5 | 4
Investigations - Other (Investigations) | 0 | 2 | 1 | 2 | 0 | 2 | 0
Inr Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hemoglobin Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 3 | 1
Ggt Increased (Investigations) | 3 | 7 | 1 | 3 | 3 | 5 | 1
Creatinine Increased (Investigations) | 5 | 10 | 14 | 18 | 9 | 8 | 6
Cholesterol High (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Cardiac Troponin T Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 7 | 3 | 4 | 3 | 6 | 2
Blood Bilirubin Increased (Investigations) | 3 | 0 | 2 | 2 | 3 | 4 | 3
White Blood Cell Decreased (Investigations) | 5 | 10 | 6 | 7 | 9 | 2 | 5
Blood Bicarbonate Decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 1 | 4 | 2 | 6 | 9 | 11
Alkaline Phosphatase Increased (Investigations) | 5 | 3 | 5 | 6 | 5 | 8 | 11
Alanine Aminotransferase Increased (Investigations) | 4 | 2 | 6 | 1 | 4 | 11 | 9
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 3 | 4 | 7 | 8 | 10 | 9
Hypokalemia (Metabolism and nutrition disorders) | 9 | 5 | 7 | 8 | 5 | 6 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 3 | 3 | 3 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 3 | 3 | 5 | 4 | 6 | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 14 | 3 | 12 | 4 | 6 | 5 | 9
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 0 | 3 | 11 | 5 | 9 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1 | 1 | 2
Glucose Intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 3 | 8 | 1 | 3 | 3 | 8
Anorexia (Metabolism and nutrition disorders) | 16 | 12 | 16 | 11 | 10 | 15 | 20
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 4 | 4 | 6 | 6
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 2 | 3 | 1 | 4
Soft Tissue Necrosis Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 2 | 0 | 3 | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 2 | 2 | 4 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 4
Muscle Weakness Trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 3
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 2
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 3 | 2 | 3 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2 | 3 | 3 | 1 | 2 | 7
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous System Disorders - Other (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 10 | 5 | 16 | 3 | 3 | 11 | 18
Paresthesia (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 5 | 5 | 9 | 2 | 2 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 5 | 5 | 6 | 5 | 2 | 8
Concentration Impairment (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Psychiatric Disorders - Other (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 3 | 2 | 6 | 8 | 4
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 5 | 2 | 1 | 2 | 2 | 1
Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 1 | 4 | 0 | 1 | 2 | 3
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Urinary Fistula (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Calculi (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 5 | 6 | 3 | 4 | 6
Urinary Incontinence (Renal and urinary disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Urinary Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 2 | 2 | 2 | 0 | 5 | 3
Glucosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 2 | 1 | 4 | 4 | 2 | 1
Cystitis Noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 1 | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 2 | 4 | 2 | 7 | 2 | 4
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 2
Uterine Hemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Perineal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 2 | 3 | 0 | 1 | 2 | 2
Vaginal Fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 3 | 0 | 0 | 0 | 5
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 5 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 7 | 1 | 0 | 2 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 8 | 6 | 13 | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 10 | 5 | 3 | 10 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3 | 0 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 9 | 1 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 3 | 5 | 6 | 6 | 3 | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 3 | 3 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 2 | 7
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail Loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 3 | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 1 | 3 | 1 | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vascular Disorders - Other (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 4 | 2 | 2 | 4 | 3 | 3
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 4 | 3 | 1 | 3 | 4
Hypertension (Vascular disorders) | 29 | 9 | 31 | 4 | 6 | 19 | 26
Hot Flashes (Vascular disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 3
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03660826/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03660826/ICF_001.pdf